CLINICAL TRIAL: NCT00075595
Title: Phase II Study of 5FU/Folinic Acid and Irinotecan as Second or Third Line Treatment in Patients With Metastatic, Unresectable, Colorectal Cancer
Brief Title: Fluorouracil, Leucovorin, and Irinotecan in Treating Patients With Recurrent or Refractory Metastatic Unresectable Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000347378; FRE-GERCOR-FOLFIRI3-C00-2; EU-20333
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Last update posted 2009-01-06 (Estimated); Status verified 2007-08

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Irinotecan; Leucovorin

INTERVENTIONS:
Drug: FOLFIRI regimen
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, leucovorin, and irinotecan, use different ways to stop tumor cells from dividing so they stop growing or die. Giving more than one chemotherapy drug may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving fluorouracil together with leucovorin and irinotecan works in treating patients with recurrent or refractory metastatic unresectable colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the time to progression and time to death from progression in patients with recurrent or refractory metastatic unresectable colorectal cancer treated with fluorouracil, leucovorin calcium, and irinotecan.

Secondary

* Determine the objective response and stabilization rate in patients treated with this regimen.
* Determine the time to treatment failure in patients treated with this regimen.
* Determine the duration of response in patients treated with this regimen.
* Determine overall survival rate in patients treated with this regimen.
* Determine the incidence of grade 3 or 4 toxicity in patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

Patients receive leucovorin calcium IV over 2 hours on day 1, irinotecan IV over 1 hour on days 1 and 3, and fluorouracil IV continuously over 46 hours beginning on day 1. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 78 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal adenocarcinoma

  * Metastatic, unresectable disease
* Meets 1 of the following criteria:

  * At least 1 unidimensionally measurable metastatic lesion at least 10 mm by spiral scan OR 20 mm by conventional scan
  * Evaluable disease
  * Evidence of disease (e.g., ascites or bone metastases) by imaging techniques
* Progressive disease as defined by 1 of the following criteria:

  * Progressive disease while receiving first-line chemotherapy
  * Recurrent disease within 6 months after completing adjuvant chemotherapy
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 to 80

Performance status

* WHO 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin < 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase < 3 times ULN

Renal

* Not specified

Cardiovascular

* No uncontrolled angina
* No myocardial infarction within the past 6 months

Gastrointestinal

* No chronic diarrhea grade 2 or greater
* No unresolved fully or partially obstructed intestine

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other underlying disease or medical condition that would preclude study participation
* No other prior malignancy except curatively treated basal cell cancer or carcinoma in situ of the cervix
* No psychological, social, familial, or geographical condition that would preclude study follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No prior irinotecan

Endocrine therapy

* Not specified

Radiotherapy

* At least 3 weeks since prior radiotherapy

Surgery

* At least 3 weeks since prior surgery

Other

* No other concurrent clinical trial participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-06

PRIMARY OUTCOMES:
Time to progression
Time to death from progression

SECONDARY OUTCOMES:
Objective response
Stabilization rate
Time to treatment failure
Duration of response
Overall survival rate
Incidence of grade 3 or 4 toxicity

CONTACTS AND LOCATIONS:
Overall Officials: May Mabro, MD — Hopital Foch
Locations (15):
- France (15):
  - Hopital Drevon, Dijon
  - Centre Hospital Universitaire Hop Huriez, Lille
  - Clinique Saint Jean, Lyon
  - Hopital Saint Joseph, Marseille
  - Intercommunal Hospital, Montfermeil
  - American Hospital of Paris, Neuilly-sur-Seine
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Bichat - Claude Bernard, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris
  - Clinique Ste - Marie, Pontoise
  - Polyclinique De Courlancy, Reims
  - Clinique Armoricaine De Radiologie, Saint-Brieuc
  - Clinique de l'Orangerie, Strasbourg
  - Centre Medico-Chirurgical Foch, Suresnes